CLINICAL TRIAL: NCT03287284
Title: Phototherapy in Association to Resistance Training in the Elderly: the Effect on Muscle Strength, Muscle Mass and Functional Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Bruno Manfredini Baroni, Phd, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 59328316.9.0000.5345
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Elderly Men
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LLLT Group (Active Comparator): Active Low Level Laser Therapy application with a dose of 240 Joules before resistance training
  Interventions: Device: Active Low Level Laser Therapy; Behavioral: Resistance Training
- Placebo Group (Placebo Comparator): Placebo Low Level Laser Therapy application before resistance training
  Interventions: Behavioral: Resistance Training; Device: Placebo Low Level Laser Therapy

INTERVENTIONS:
Device: Active Low Level Laser Therapy — Active application of Low Level Laser Therapy with a dose of 240 Joules
  Arms: LLLT Group
Behavioral: Resistance Training — Resistance Training
Device: Placebo Low Level Laser Therapy — Placebo application of Low Level Laser Therapy
  Arms: Placebo Group

SUMMARY:
Phototherapy has been largely used in rehabilitation programs due to its analgesic, antiinflammatory and healing effects. Lately, its effects of optimizing the results of resistance training on young individuals have been studied. However, there is a lack of studies on its effect on the elderly population. The objective of the present study is to verify the effect of Low-Level Laser Therapy (LLLT) on the results of resistance training in the elderly. The study will be a randomized doubled-blinded controlled trial. 30 elderly men with age ranging from 60 to 80 years will be included and randomized between Placebo Group (placebo LLLT + Resistance Training) and LLLT Group (active LLLT + Resistance Training). All volunteers will be submitted to a control period of four weeks before the beginning of the resistance training, which will have 12 weeks of duration. The assessments will be done at baseline, after the control period and after the training period. The training sessions will be performed twice a week and the training protocol will be performed with repetition maximum periodization. The LLLT will be applied before the training sessions on eight points of the quadriceps muscles, leading to a total of 240 Joules on each leg. The placebo LLLT will be applied on the same way, but with the equipment turned off. The assessments will include muscle architecture by ultrasonography, muscle strength by isokinetic dynamometer and 1 Repetition Maximum test of leg-extension and leg-press exercises, and functional capacity by the 6-Minute Walking Test, 30s Sit to Stand Test, Timed Up-and-Go Test and Stair Ascent Test.

ELIGIBILITY:
Inclusion Criteria:

* Elderly men with age ranging from 60 to 80 years in condition to participate in the strength training program.

Exclusion Criteria:

* Individuals who already participate in strength training programs;
* Individuals who participated in strength training programs less than three months before the beginning of the study;
* Individuals with any kind musculoskeletal injuries in the lower limbs that impair the performance of the exercises;
* Individuals with contraindications to the performance of high intensity exercises, such as cardiovascular or neurological diseases;
* Individuals with difficulties in understanding and/or performing the exercises;
* Individuals who did not attend to at least 85% of the sessions or had 02 consecutive absences and did not recover them.

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Isokinetic peak torque of quadriceps muscle | Change from baseline in isokinetic peak torque at 12 weeks

SECONDARY OUTCOMES:
Leg-extension 1RM test | Change from baseline in leg-extension 1RM test at 12 weeks
Leg-press 1RM test | Change from baseline in leg-press 1RM test at 12 weeks
Muscle architecture | Change from baseline in muscle architecture at 12 weeks
Physical Function | Change from baseline in physical function at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Sul, Pôrto Alegre, Brazil